CLINICAL TRIAL: NCT02833311
Title: Examining the Usability of Computer Tablets to Promote Symptom Self-management and Engagement in Healthy Behaviors in Adults With Chronic Conditions
Brief Title: e-Mobile Tablet for People With Chronic Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Matthew Plow, Assistant Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12-14-25
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Results first posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2022-07

CONDITIONS: Fibromyalgia; Multiple Sclerosis; Osteoarthritis; Sjögren's Syndrome; Parkinson's Disease
Keywords: Neuromusculoskeletal condition
MeSH Terms: conditions — Fibromyalgia; Multiple Sclerosis; Osteoarthritis; Sjogren's Syndrome; Parkinson Disease | interventions — Paper

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Computer Tablet Group (Active Comparator): Participants will first meet once with a trained health education specialist. During this meeting the health education specialist will work with the participant in setting constructive and manageable goals and how to achieve them safely. Participants will then receive weekly follow-up phone calls to discuss progression and/or possible trouble-shooting strategies. Participants will be asked to set goals related to increasing self managing health behaviors. Participants will be encouraged to self-monitor goals, behaviors and symptoms using a computer tablet.
  Interventions: Behavioral: Computer Tablet Group
- Paper and Pencil Group (Active Comparator): Participants will first meet once with a trained health education specialist. During this meeting the health education specialist will work with the participant in setting constructive and manageable goals and how to achieve them safely. Participants will then receive weekly follow-up phone calls to discuss progression and/or possible trouble-shooting strategies. Participants will be asked to set goals related to increasing self managing health behaviors. Participants will be encouraged to self-monitor goals, behaviors and symptoms using a paper-pencil diary.
  Interventions: Behavioral: Paper and Pencil Group
- Contact Control Group (Active Comparator): Participants will first meet once with a health education specialist. During this meeting the health education specialist will provide general information about engaging in healthy behaviors. Information will primarily focus on the benefits of engaging in healthy behaviors and safety precautions. Participants will then receive weekly follow-up phone calls to discuss various health topics.
  Interventions: Behavioral: Contact Control Group

INTERVENTIONS:
Behavioral: Computer Tablet Group — A computer tablet application to set goals,self-monitor healthy behaviors, record condition-related symptom impact, and self-manage a problematic symptom.
  Arms: Computer Tablet Group
Behavioral: Paper and Pencil Group — Use of paper and pencil diaries and worksheets to set goals, record condition-related symptom impact, and self-monitor behaviors.
  Arms: Paper and Pencil Group
Behavioral: Contact Control Group — Participants are prescribed an exercise program and given information on healthy eating.
  Arms: Contact Control Group

SUMMARY:
Maintaining a healthy diet and engaging in routine physical activity may help decrease severity of symptoms, prevent secondary conditions, and slow functional decline in people with disabling neuromusculoskeletal conditions. However, people with these conditions face many health barriers to engaging in healthy behaviors. With the advent of portable technologies, such as smart phones, tablets and PDAs, there is a need to explore whether these technologies can help people with disabling conditions to stay motivated and overcome barriers to engaging in healthy behaviors.

DETAILED DESCRIPTION:
The overarching goal of this mixed methods, comparative effectiveness randomized controlled pilot study is to evaluate whether goal setting, self-monitoring, and barrier management using a computer tablet can increase physical activity behavior, improve nutritional habits, and promote health-related quality of life in people with disabling neuromusculoskeletal conditions. Our hypothesis is that, in comparison to the standard care contact control group, participants in both the tablet group and the paper and pencil group will yield significant improvements in healthy behaviors,with the tablet group yielding significantly larger increases.

ELIGIBILITY:
Inclusion Criteria:

* Physician-confirmed diagnosis of a neuro-musculoskeletal condition or disease of the nerves, muscles, and/or bones that results in functional limitations
* Physician consent to engage in home exercise/physical activity program
* Regularly inactive (i.e., engaging in 90 minutes or less of purposeful physical activity each week)
* Scoring ≤17 mental composite and ≤16 physical composite on the Global Health Questionnaire.
* Have internet access (i.e., home, library or other WiFi location)

Exclusion Criteria:

* If the only disabling condition reported is not considered a neuro-musculoskeletal disease
* Have hand-motor function impairments that would limit use of the tablet
* Often engage in healthy eating habits
* Are frequent fallers (i.e., more than 3 falls per month)
* Have a diagnoses of chronic obstructive pulmonary disease, serious mental health disorder, chronic heart failure, myocardial infarction, and other unstable/severe cardiovascular conditions, and uncontrolled diabetes mellitus (e.g., admission to the hospital within the past 6 months for uncontrolled diabetes)
* Have severe cognitive deficits
* Reports consistently tracking and monitoring health behaviors
* Unable to effectively use the tablet technology during the pre-intervention usability demonstration

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A Plow, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Plow M, Golding M. Using mHealth Technology in a Self-Management Intervention to Promote Physical Activity Among Adults With Chronic Disabling Conditions: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2017 Dec 1;5(12):e185. doi: 10.2196/mhealth.6394. PMID 29196279

RESULTS

PARTICIPANT FLOW:
Groups:
- Computer Tablet Group: A computer tablet application to set goals,self-monitor healthy behaviors, record condition-related symptom impact, and self-manage a problematic symptom.
  Computer Tablet Group: Participants will first meet once with a trained health education specialist. During this meeting the health education specialist will work with the participant in setting constructive and manageable goals and how to achieve them safely. Participants will then receive weekly follow-up phone calls to discuss progression and/or possible trouble-shooting strategies. Participants will be asked to set goals related to increasing self managing health behaviors. Participants will be encouraged to self-monitor goals, behaviors and symptoms using a computer tablet.
- Paper and Pencil Group: Use of paper and pencil diaries and worksheets to set goals, record condition-related symptom impact, and self-monitor behaviors.
  Paper and Pencil Group: Participants will first meet once with a trained health education specialist. During this meeting the health education specialist will work with the participant in setting constructive and manageable goals and how to achieve them safely. Participants will then receive weekly follow-up phone calls to discuss progression and/or possible trouble-shooting strategies. Participants will be asked to set goals related to increasing self managing health behaviors. Participants will be encouraged to self-monitor goals, behaviors and symptoms using a paper-pencil diary.
- Standard Treatment Control Group: Participants are prescribed an exercise program and given information on healthy eating.
  Standard Treatment Control Group: Participants will first meet once with a health education specialist. During this meeting the health education specialist will provide general information about engaging in healthy behaviors. Information will primarily focus on the benefits of engaging in healthy behaviors and safety precautions. Participants will then receive weekly follow-up phone calls to discuss various health topics.
Period: Overall Study
Arm/Group | Computer Tablet Group | Paper and Pencil Group | Standard Treatment Control Group
Started | 15 | 16 | 15
Completed | 13 | 15 | 15
Not Completed | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Computer Tablet Group | Paper and Pencil Group | Standard Treatment Control Group | Total
Number analyzed (Participants) | 15 | 16 | 15 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 11 | 11 | 36
  >=65 years | 1 | 5 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.93 (5.52) | 59.38 (10.2) | 55 (11.58) | 57.8 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 12 | 39
  Male | 2 | 2 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 15 | 46

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline in Physical Activity
Description: Physical Activity and Disability Survey-Revised was administered to assess physical activity behavior. Scores can range from -2.7493 to 3.3671. Higher scores on the Physical Activity and Disability Survey-Revised indicates increased physical activity levels.
Time Frame: Outcomes were administered immediately before the intervention and again 6-weeks later
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Contact Control Group: Participants are prescribed an exercise program and given information on healthy eating.
  Standard Treatment Control Group: Participants will first meet once with a health education specialist. During this meeting the health education specialist will provide general information about engaging in healthy behaviors. Information will primarily focus on the benefits of engaging in healthy behaviors and safety precautions. Participants will then receive weekly follow-up phone calls to discuss various health topics.
Arm/Group | Computer Tablet Group | Paper and Pencil Group | Contact Control Group
Number analyzed (Participants) | 13 | 15 | 15
units on a scale
  Pretest | 0.36 (0.77) | 0.31 (1.01) | 0.43 (0.68)
  Posttest | 0.76 (0.92) | 0.55 (1.15) | 0.36 (0.61)

2. Secondary Outcome: Changes From Baseline in Self-Report Physical Function
Description: Patient Reported Outcome Measurement information System (PROMIS) Physical Function (PF) was used to measure self-report physical function. Measures are scored on a T-score metric. High scores indicate more of the concept being measured. A score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population.
Time Frame: Outcomes were administered immediately before the intervention and again 6-weeks later
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Computer Tablet Group | Paper and Pencil Group | Contact Control Group
Number analyzed (Participants) | 13 | 15 | 15
units on a scale
  Pretest | 39.87 (5.87) | 38.89 (3.14) | 42.44 (5.45)
  Posttest | 38.44 (7.54) | 37.91 (4.52) | 41.51 (3.96)

3. Secondary Outcome: Changes From Baseline in 6-minute Walking Test
Time Frame: Outcomes were administered immediately before the intervention and again 6-weeks later
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Computer Tablet Group | Paper and Pencil Group | Contact Control Group
Number analyzed (Participants) | 13 | 15 | 15
meters
  Pretest | 303.69 (87.23) | 316.32 (117.58) | 362.32 (91.01)
  Posttest | 327.46 (68.32) | 320.61 (122.02) | 385.23 (82.26)

4. Secondary Outcome: Changes From Baseline in Self-Efficacy
Description: Exercise Confidence Survey was used to measure self-efficacy. The survey asks about confidence in sticking to an exercise program and making time for exercise. This is a 12 item questionnaire and scores ranges from 1 to 60. A higher score indicates increased confidence to engage in exercise.
Time Frame: Outcomes were administered immediately before the intervention and again 6-weeks later
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Computer Tablet Group | Paper and Pencil Group | Contact Control Group
Number analyzed (Participants) | 13 | 15 | 15
units on a scale
  Pretest | 3.26 (0.96) | 3.29 (0.91) | 3.33 (0.45)
  Posttest | 3.25 (0.82) | 3.42 (0.76) | 2.97 (0.55)

5. Secondary Outcome: Changes From Baseline in Weight
Time Frame: Outcomes were administered immediately before the intervention and again 6-weeks later
Population: 3 participants (2 in the computer tablet group and 1 in the paper and pencil group) were missing weight data for posttest timepoint. These participants were removed from analysis.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Computer Tablet Group | Paper and Pencil Group | Contact Control Group
Number analyzed (Participants) | 13 | 15 | 15
kg
  Pretest | 91.78 (28.50) | 88.80 (22.12) | 81.71 (22.64)
  Posttest | 91.32 (27.97) | 87.58 (20.12) | 81.56 (23.05)

ADVERSE EVENTS:
Arm/Group | Computer Tablet Group | Paper and Pencil Group | Standard Treatment Control Group
Serious Adverse Events (participants affected / at risk) | 3/15 | 3/16 | 1/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Computer Tablet Group (N=15) | Paper and Pencil Group (N=16) | Standard Treatment Control Group (N=15)
Falls (General disorders) | 3 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No